CLINICAL TRIAL: NCT06724952
Title: Clinical Study Evaluating Anti Rheumatic Activity and The Role of Silymarin in Attenuating Methotrexate Toxicity in Patients With Rheumatoid Arthritis
Brief Title: Effect of Silymarin in Rheumatoid Arthritis Patients Treated With Methotrexate
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Hend Mohsen Mohamed El-metwally, Teaching Assistant in clinical pharmacy at Horus University and master degree student, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Effect of Silymarin in RA
Record Dates: First submitted 2024-10-06; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: Rheumatoid Arthritis; Silymarin; Methotrexate
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Silymarin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- MTX S.C or IM _ Silymarin tab (Active Comparator): IM or S.C MTX plus Silymarin 140 mg Tab once daily
  Interventions: Drug: MTX S.C or IM and Silymarin 140 mg tab
- MTX S.C or IM _ Placebo tablet (Placebo Comparator): IM or S.C MTX plus Placebo Tablet once daily
  Interventions: Drug: MTX S.C or IM

INTERVENTIONS:
Drug: MTX S.C or IM and Silymarin 140 mg tab — IM or S.C Methotrexate plus Silymarin tablets 140 mg once daily for 3 months.
  Arms: MTX S.C or IM _ Silymarin tab
Drug: MTX S.C or IM — IM or SC Methotrexate plus placebo tablet once daily for 3 months.
  Arms: MTX S.C or IM _ Placebo tablet

SUMMARY:
The goal of this clinical trial is to evaluate the anti-rheumatic activity and the role of silymarin in attenuating methotrexate toxicity in patients with rheumatoid arthritis.

Methodology:

This is a randomized, double blind placebo controlled parallel study that will be conducted on 44 patients with active rheumatoid arthritis.

Group1 (placebo group; n=22) which will receive IM or SC Methotrexate plus placebo tablet once daily for 3 months.

Group2 (Silymarin group; n=22) which will receive IM or SC Methotrexate plus Silymarin tablets 140 mg once daily for 3 months.

Duration: 3 months

Monitoring:

Participants will be followed up by weekly telephone calls and monthly direct meeting at scheduled visits to assess their adherence and to report any drug related adverse effects.

In summary, this clinical trial is designed to determine if Silymarin is a safe and effective treatment for Rheumatoid Arthritis Patients Treated with Methotrexate by comparing its effects to a placebo and closely monitoring participants throughout the study.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is an autoimmune disorder in which immune systems mistakenly attacks the host body systems. Its clinical features are often characterized as chronic synovial non-infectious inflammation, cartilage, and bone destruction (1). Currently, no effective drugs can be used to cure RA in the clinic. For the treatment of RA, recommended medications include disease-modifying anti-rheumatic drugs (DMARDs) and biologic agents, which intend to achieve the remission of symptoms, but these medications also confer severe side effects when they exert therapeutic efficiency (2). Due to drug resistance and side effects, a big proportion of RA patients do not effectively respond to the treatment and urgently need new drugs or therapeutic strategies.

Approximate 60% of RA patients are overweight and suffering from metabolic disorders (3). Clinical features of lipid paradox often occur in active RA patients, leading to high risk of developing cardiovascular morbidity and mortality (4-6). In addition, the deregulated lipid metabolism is yet present in the early stage of RA and/or pre-RA (7). In recent years, lipid-lowering therapy with statins is demonstrated to be effective in RA treatment (8,9) and in the prevention of the dyslipidemia development in RA patients (10). In short, we can confirm that lipid metabolism must be implicated in the pathogenesis of RA, which conserves the drug-target capacity for therapeutic discovery against RA in the clinic, especially for overweight patients with dyslipidemia (10).

Silymarin, a major flavonoid from milk thistle (silymarin), has been used to treat many liver disorders, such as nonalcoholic steatohepatitis (NASH), cirrhosis, and liver cancer, based on its anti-oxidant, anti-inflammation, anti-fibro genetic and lipid-lowering pharmacological activities (11).

Overexpression of liver X receptor α (LXRα) and several key lipogenic enzymes regulated by LXRα, including lipoprotein lipase (LPL), cholesterol 7α and 27α hydroxylase (CYP7A, CYP27A), adipocyte fatty acid-binding protein (aP2/FABP4) and fatty acid translocase (CD36/FAT), were observed in AIA rats, which mostly accounted for dyslipidemia during arthritis development. Metabolomics, docking technology, and biochemical results indicated that antiarthritis effects of silymarin related to suppressing the up-regulated LXRα and abnormal lipid metabolism. Notably, activation of LXRα could potentiate cell inflammatory process induced by LPS (Lipopolysaccharide) through the regulation of NF-κB pathway, however, suppression of LXRα agonism by siRNA or silymarin reduced the nuclear translocation of NF-κB as well as the induction of downstream cytokines, indicating LXRα agonism is the important factor for the arthritis development and could be a potential target (12). Considering the priority of silymarin in drug-safety, and the potential in improving lipid metabolism, therefore our effort attempted to explore the therapeutic potential of silymarin against RA with dyslipidemia, effect of silymarin on lipid profile and lipoprotein lipase and decipher associated molecular mechanisms accordingly.

Methotrexate has remained the "anchor drug" for most patients since the late 1980s (13). However, despite its long-term and widespread use for RA, methotrexate induce liver and nephrotoxicity, In study done by Adel A Hagag et al, on 80 children with newly diagnosed Acute Lymphoblastic Leukemia (ALL) received Silymarin 420 mg/day in 3 divided doses for one week after each MTX dose indicate that Silymarin improved some hepatic and renal functions in children with ALL who received MTX-based chemotherapy protocols (14).

In the present study, we evaluate the lipid profile and the major lipid metabolic enzymes in rheumatoid arthritis patients treated with methotrexate, and further explore the effects of silymarin in ameliorating both arthritis, dyslipidemia, the underlying mechanism of silymarin against RA through the regulation of lipoprotein lipase / lipid metabolism as well as effect of silymarin on methotrexate liver and renal toxicity.

ELIGIBILITY:
* Inclusion criteria:

  * Patients with active rheumatoid arthritis (not in remission) according to 28 joints disease activity score (DAS-28) >2.6.
  * Age range between 18 and 60 years old.
  * Both sexes.
  * Sex ratio, age, disease activity, and disease duration matched patients.
  * Patients receive methotrexate plus traditional therapy
* Exclusion criteria:

  * Patients with renal or hepatic diseases (chronic liver disease, liver cirrhosis, alcoholic hepatitis, or chronic alcoholism).
  * Patients receiving biological DMARDs.
  * Patients with hypersensitivity to study medications.
  * Patients using antioxidants except silymarin.
  * Pregnant and lactating females.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-12-10 (Estimated); Primary Completion 2025-03-10 (Estimated); Study Completion 2025-04-10 (Estimated)

PRIMARY OUTCOMES:
Calculation of DAS-28-CRP score for measure disease activity. | From enrollment to the end of treatment at 3 months
  This is a score for measure of disease activity in Rheumatoid Arthritis; Less than 2.6 mean RA is in remission, 2.6 to 3.2 mean low level of disease activity, More than 3.2 mean active disease that may require change in medication, More than 5.1 mean very active disease that requires careful monitoring and adjustment to medication

SECONDARY OUTCOMES:
Measurement of serum Nuclear factor kappa-B p65 (NF-κ B p65) & Lipoprotein lipase (LPL). | From enrollment to the end of treatment at 3 months
  Before and 3 months after the intervention, 5 ml of venous blood will be withdrawn by antecubital venipuncture from each participant between 8:30 and 10:30 am. Blood samples will be transferred into a plain test tube and centrifuged at 3000 rpm for 10 min. the separated serum will be used for determination of: serum Nuclear factor kappa-B p65 (NF-κ B p65) & Lipoprotein lipase (LPL).
  serum Nuclear factor kappa-B p65 (NF-κ B p65): one of the main inflammatory pathways in the Autoimmune Disease (AD) Rheumatoid Arthritis (RA), which exhibits high levels of inflammatory cytokines such as IL-1, TNFa and IL-6.
  Lipoprotein lipase: Overexpression of liver X receptor α (LXRα) and several key lipogenic enzymes regulated by LXRα, including lipoprotein lipase (LPL) were observed in adjuvant-induced arthritis.

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Internal Medicine, Rheumatology and Immunology Department, Mansoura University Hospital, Mansoura, 35511, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hagag AA, Elgamsy MA, El-Asy HM, Mabrouk MM. Protective Role of Silymarin on Hepatic and Renal Toxicity Induced by MTX Based Chemotherapy in Children with Acute Lymphoblastic Leukemia. Mediterr J Hematol Infect Dis. 2016 Sep 1;8(1):e2016043. doi: 10.4084/MJHID.2016.043. eCollection 2016. PMID 27648206
- [Result] Weinblatt ME, Coblyn JS, Fox DA, Fraser PA, Holdsworth DE, Glass DN, Trentham DE. Efficacy of low-dose methotrexate in rheumatoid arthritis. N Engl J Med. 1985 Mar 28;312(13):818-22. doi: 10.1056/NEJM198503283121303. PMID 3883172
- [Result] Xie Y, Feng SL, Mai CT, Zheng YF, Wang H, Liu ZQ, Zhou H, Liu L. Suppression of up-regulated LXRalpha by silybin ameliorates experimental rheumatoid arthritis and abnormal lipid metabolism. Phytomedicine. 2021 Jan;80:153339. doi: 10.1016/j.phymed.2020.153339. Epub 2020 Sep 19. PMID 33038868
- [Result] Karimi G, Vahabzadeh M, Lari P, Rashedinia M, Moshiri M. "Silymarin", a promising pharmacological agent for treatment of diseases. Iran J Basic Med Sci. 2011 Jul;14(4):308-17. PMID 23492971
- [Result] Nurmohamed MT, Dijkmans BA. Dyslipidaemia, statins and rheumatoid arthritis. Ann Rheum Dis. 2009 Apr;68(4):453-5. doi: 10.1136/ard.2008.104497. No abstract available. PMID 19286903
- [Result] Soulaidopoulos S, Nikiphorou E, Dimitroulas T, Kitas GD. The Role of Statins in Disease Modification and Cardiovascular Risk in Rheumatoid Arthritis. Front Med (Lausanne). 2018 Feb 8;5:24. doi: 10.3389/fmed.2018.00024. eCollection 2018. PMID 29473041
- [Result] Das S, Mohanty M, Padhan P. Outcome of rheumatoid arthritis following adjunct statin therapy. Indian J Pharmacol. 2015 Nov-Dec;47(6):605-9. doi: 10.4103/0253-7613.169585. PMID 26729950
- [Result] Kerekes G, Nurmohamed MT, Gonzalez-Gay MA, Seres I, Paragh G, Kardos Z, Barath Z, Tamasi L, Soltesz P, Szekanecz Z. Rheumatoid arthritis and metabolic syndrome. Nat Rev Rheumatol. 2014 Nov;10(11):691-6. doi: 10.1038/nrrheum.2014.121. Epub 2014 Aug 5. PMID 25090948
- [Result] Giles JT, Allison M, Blumenthal RS, Post W, Gelber AC, Petri M, Tracy R, Szklo M, Bathon JM. Abdominal adiposity in rheumatoid arthritis: association with cardiometabolic risk factors and disease characteristics. Arthritis Rheum. 2010 Nov;62(11):3173-82. doi: 10.1002/art.27629. PMID 20589684
- [Result] Erum U, Ahsan T, Khowaja D. Lipid abnormalities in patients with Rheumatoid Arthritis. Pak J Med Sci. 2017 Jan-Feb;33(1):227-230. doi: 10.12669/pjms.331.11699. PMID 28367205
- [Result] Amezaga Urruela M, Suarez-Almazor ME. Lipid paradox in rheumatoid arthritis: changes with rheumatoid arthritis therapies. Curr Rheumatol Rep. 2012 Oct;14(5):428-37. doi: 10.1007/s11926-012-0269-z. PMID 22802154
- [Result] Roubenoff R, Roubenoff RA, Cannon JG, Kehayias JJ, Zhuang H, Dawson-Hughes B, Dinarello CA, Rosenberg IH. Rheumatoid cachexia: cytokine-driven hypermetabolism accompanying reduced body cell mass in chronic inflammation. J Clin Invest. 1994 Jun;93(6):2379-86. doi: 10.1172/JCI117244. PMID 8200971
- [Result] Guo Q, Wang Y, Xu D, Nossent J, Pavlos NJ, Xu J. Rheumatoid arthritis: pathological mechanisms and modern pharmacologic therapies. Bone Res. 2018 Apr 27;6:15. doi: 10.1038/s41413-018-0016-9. eCollection 2018. PMID 29736302
- [Result] McInnes IB, Schett G. The pathogenesis of rheumatoid arthritis. N Engl J Med. 2011 Dec 8;365(23):2205-19. doi: 10.1056/NEJMra1004965. No abstract available. PMID 22150039